CLINICAL TRIAL: NCT02151669
Title: EFFECT OF A MEDITERRANEAN DIET INTERVENTION IN PULMONARY FUNCTION IN SMOKERS: A MULTICENTER RANDOMIZED CLINICAL TRIAL IN PRIMARY CARE CENTERS
Brief Title: Diet Intervention Spirometry and Tobacco
Acronym: DIET
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fundacio d'Investigacio en Atencio Primaria Jordi Gol i Gurina (Other)
Collaborators: Preventive Services and Health Promotion Research Network (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 4R13/068
Record Dates: First submitted 2014-05-26; First posted 2014-05-30 (Estimated); Last update posted 2023-02-27 (Actual); Status verified 2023-02

CONDITIONS: Pulmonary Function
Keywords: Mediterranean diet; Smoking/tobacco; Spirometry
MeSH Terms: conditions — Smoking | interventions — Diet, Mediterranean

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Mediterranean Diet Group (Experimental): Nutritional intervention to enhance the traditional Mediterranean diet pattern using new technology as an educational tool in primary care: DIET blog. Participants will be referred to a single annual visit and one group session per year for two years.
  Interventions: Behavioral: Mediterranean Diet
- Control group (No Intervention): Participants of control group will be referred to your doctor or nurse with reference to a report on specific according to your personal situation dietary recommendations.

INTERVENTIONS:
Behavioral: Mediterranean Diet — Nutritional intervention conducted by a dietitian who designs a nutrition program to enhance the traditional Mediterranean diet pattern using new technology as an educational tool in primary care: DIET blog. Participants will be referred to a single annual visit and one group session per year for two years.
  Arms: Mediterranean Diet Group

SUMMARY:
Epidemiologic studies suggest that some nutrients can be affected lung function. Moreover, no previous studies have prospectively evaluated the effect of the Mediterranean dietary pattern in lung function in smokers. Phase II of the RESET study , a clinical trial to evaluate the efficacy of a motivational smoking intervention based on information obtained by spirometry (FIS project PI11/01962).

DETAILED DESCRIPTION:
Design: Multicenter randomized controlled trial in primary care. Sample: We will recruit 80 smokers from 35 to 70 years without history of lung disease. Subjects will be randomly assigned to control or intervention group (1:1).

Study variables: We measure socio-demographic, clinical, anthropometry and spirometry data. Food consumption will be evaluated by a semi-quantitative food frequency questionnaire (FFQ), energy expenditure in physical activity by the Minnesota Leisure Time Activity questionnaire and adherence to Mediterranean Diet by a 14-item questionnaire.

Intervention: Nutritional intervention conducted by a dietitian who designs a nutrition program to enhance the traditional Mediterranean diet pattern using new technology as an educational tool in primary care: DIET blog. Participants will be referred to a single annual visit and one group session per year for two years.

Analysis: All analyses will be based on intention-to-treat. The results will be considered clinically relevant when it detects a difference in lung function (decreased FEV1) >10-12 ml/year. A p-value of <0.05 will defined statistical significance.

ELIGIBILITY:
Inclusion Criteria:

* Being active smokers at the time of enrollment with an cumulative consumption more than 10 packs / year
* Having Internet access and regular use of new technologies in general or have help for it.
* Having participated in the first phase of the project: RESET study (PI11/01962).

Exclusion Criteria:

* Any evidence of previous diagnosis of respiratory disease,
* Suffering from a terminal or chronic disorder that alters the baseline parameters or hinder the completion of testing and required test during the study period,
* Inability to track for any reason,
* Express refusal of the patient to continue in the study

Ages: 35 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2013-11; Primary Completion 2015-05 (Actual); Study Completion 2016-11 (Actual)

PRIMARY OUTCOMES:
Changes in lung function | 2 years
  Assess the relationship between lung function and adherence to a Mediterranean Diet and its components

SECONDARY OUTCOMES:
Lung function and anthropometric parameters | 2 years
  Assess the relationship between lung function and anthropometric parameters such as waist circumference and BMI.
Lung function and effectiveness of a nutritional educational tool 2.0 | 2 years
  To evaluate the effectiveness of using an nutritional educational tool 2.0 to increase adherence to a Mediterranean diet: blog.

CONTACTS AND LOCATIONS:
Overall Officials: Francisco Martín Luján, MD, Principal Investigator — Catalan Institute of Health
Locations (1):
- Unitat de Recerca. CAP Sant Pere, Reus, Tarragona, Spain

REFERENCES:
- [Result] Salamanca-Gonzalez P, Valls-Zamora RM, Pedret-Figuerola A, Sorli-Aguilar M, Santigosa-Ayala A, Catalin RE, Palleja-Millan M, Sola-Alberich R, Martin-Lujan F, The Cenit Research Group Investigators. Effectiveness of a Motivational Nutritional Intervention through Social Networks 2.0 to Increase Adherence to the Mediterranean Diet and Improve Lung Function in Active Smokers: The DIET Study, a Randomized, Controlled and Parallel Clinical Trial in Primary Care. Nutrients. 2021 Oct 14;13(10):3597. doi: 10.3390/nu13103597. PMID 34684600
- [Result] Sorli-Aguilar M, Martin-Lujan F, Flores-Mateo G, Arija-Val V, Basora-Gallisa J, Sola-Alberich R; RESET Study Group investigators. Dietary patterns are associated with lung function among Spanish smokers without respiratory disease. BMC Pulm Med. 2016 Nov 25;16(1):162. doi: 10.1186/s12890-016-0326-x. PMID 27884188
- [Derived] Sorli-Aguilar M, Martin-Lujan F, Santigosa-Ayala A, Pinol-Moreso JL, Flores-Mateo G, Basora-Gallisa J, Arija-Val V, Sola-Alberich R. Effects of mediterranean diet on lung function in smokers: a randomised, parallel and controlled protocol. BMC Public Health. 2015 Jan 31;15:74. doi: 10.1186/s12889-015-1450-x. PMID 25636808